CLINICAL TRIAL: NCT07180030
Title: Determination of Reliability, Validity, and Minimal Detectable Change (MDC) of the Figure-of-eight Backward Walking Test in Elderly Adults
Brief Title: Figure-of-eight Backward Walk Test in Elderly
Acronym: elderly
Status: Recruiting | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Associate Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: figure-of-eight backward walk
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Elderly (People Aged 65 or More); Balance; Dynamic Balance; Backward Walking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/study group: Healthy elderly individuals over the age of 65 living in the city center of Kahramanmaraş

SUMMARY:
Mobility is a fundamental element of healthy aging. Balance is a necessary function during mobility for all movements throughout life in elderly individuals. Falls due to balance disorders in elderly individuals cause a decrease in the quality of life. Studies in the literature indicate that 13% of individuals aged 65-69 experience falls, and this rate rises to 46% in individuals over 85. Lower extremity muscle volume and strength gradually decrease with aging. This decreased muscle strength directly impacts individuals' activities of daily living.Normal walking speed for elderly individuals is related to balance and overall health performance. However, walking assessments generally focus on walking activities in a forward direction and in a straight line. However, in daily life, we may need to sit on a chair, walk backward to navigate a narrow space, or change direction suddenly due to obstacles or environmental cues. Walking backward requires more complex motor control, and these gait training programs are known to be effective in improving balance and walking skills.Clinically, balance assessments in the elderly persons are commonly measured by using the TUG, 10-meter walk test, functional reach test, 4-square step test, and Berg balance scale. The methods used to assess balance are still not fully standardized. The best test for assessing dynamic balance and fall risk is still up for debate, especially when it comes to elderly individuals who live freely in the community. Further research is needed to determine whether lateral walking tests can identify those at high risk of falling in elderly adults. The purpose of this study was to determine the reliability, validity, and minimal detectable change (MDC) of the Figure-of-8 backward walking test in healthy elderly adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy elderly individuals over 65 years of age.
* Elderly individuals who have fluent in Turkish and able to communicate.
* Elderly individuals who have no cognitive impairment.

Exclusion Criteria:

* Elderly individuals who have any neurological problems (Parkinson's, hemiplegia, etc.)
* Elderly individuals who have any orthopedic problems (fractures, etc., in the last year)
* Elderly individuals who have a body mass index (BMI) ≥ 40 kg/m2
* Elderly individuals who havevision problems
* Elderly individuals who have had any lower extremity surgery in the last year
* Elderly individuals who use any mobility aids
* Elderly individuals who refuse to participate in the study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: It is planned to include elderly individuals over 65 years of age residing in the Kahramanmaraş city center in the scope of the research, and healthy elderly individuals over 65 years of age (n=87) who can be reached by random sampling method will be included in the research.
Sampling Method: Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
figure-of-eight backward walking test | On the day 1, in the first session, the first assessor (PT1) will perform the F8BWT twice. In the second session, the second assessor (PT2) will perform the F8BWT twice.
  In the figure-of-eight backward walking (F8BWT) test, participants begin at the midpoint of two cones 1.5 m apart. Participants walk backward, circle both cones, and record the time it takes to return to the starting point. The test is administered by both raters on the first and second days.The assessments will be conducted by two separate specialists(physiotherapists). Individuals' completion times for each activity during the tests will be recorded using a stopwatch. Assessments will be conducted over two days, in two sessions per day. On the first day, in the first session, the first assessor (PT1) will perform the F8BWT twice. In the second session, the second assessor (PT2) will perform the F8BWT twice. The average of the two recorded times will be noted. On the second day of the assessment, the PT2 will begin by performing the F8BWT. PT2 will then perform the F8BWT twice. The average of the two recorded times will be noted.

SECONDARY OUTCOMES:
SOCIODEMOGRAPHIC FORM | On the day1, in the first session, the first assessor (PT1) will record.
  Demographic information (age, height, weight, gender, education level, medication use, chronic diseases, medications), history and number of falls in the last year, and history of surgery on the lower extremity will be questioned.
8-Figure Walk Test | On the day1, in the first session, the first assessor (PT1) will record.
  This test is used to evaluate individuals' walking and balance performance. In the figure-of-eight backward walking test, participants start from the midpoint of two cones 1.5 m apart. Participants walk forward, circle each cone, and record the time it takes to return to the starting point.
Timed Up and Go Test (TUG) | On the first day1, in the first session, the first assessor (PT1) will record.
  In the timed up and go test, the time required for the participant to rise from a chair, walk 3 m, turn, walk back, and sit back in the chair is recorded. Participants are asked to remove their shoes if they have any that might affect walking performance.
Modified 4-Square Step Test (mFSST) | On the first day1, in the first session, the first assessor (PT1) will record.
  The mFSST is a dynamic balance test that involves forward, backward, and sideways steps. A square is drawn on the floor and consists of four equal parts. These are numbered clockwise, 1-2-3-4. Subjects are asked to complete the test one step at a time, following the command "Start," 1-2-3-4, and then 4-3-2-1, without scraping their feet. The elapsed time is recorded.
3-Meter Backward Walk Test (3MGYT) | On the day1, in the first session, the first assessor (PT1) will record.
  For this test, a 3-meter distance is marked with a tape, and participants are asked to walk backwards, with their heels on the tape. During the test, participants are asked to walk as fast as possible, but running is not allowed. Participants may look back if they wish. The time is measured and recorded.
Tandem Test | On the day1, in the first session, the first assessor (PT1) will record.
  This test, used to assess balance, is administered with eyes open and eyes closed, alternating between each foot. The participant is asked to stand with one foot in front of the other (tandem stance), first with eyes open, then with eyes closed, for 10 seconds. They are asked to place the foot they find most comfortable with either forward or backward. The times during the test are recorded in seconds using a stopwatch.
One-Legged Standing Test | On the day1, in the first session, the first assessor (PT1) will record.
  In the one-leg standing test, participants are asked to stand on one foot of their choice while lifting the other foot, keeping it away from the ground and other body parts. If the foot touches the ground or the extremity in contact with the ground changes position during the test, the test is terminated and the time is recorded. Alternatively, if participants can stand on one foot for 30 seconds, the test is terminated and the time is recorded.
The Falls Efficacy Scale-International (FES-I) | On the day1, in the first session, the first assessor (PT1) will record.
  The The Falls Efficacy Scale-International (FES-I) is a questionnaire developed to assess the tendency to fall during activities of daily living. The test has a 4-point Likert-type scale (1- not at all concerned, 2- somewhat concerned, 3- quite concerned, and 4- very concerned). The 16-item questionnaire requires a minimum score of 16 and a maximum score of 64. Increasing scores indicate deterioration of balance (23). Participants complete the FES-I questionnaire in a quiet environment, and the score is then calculated.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel tat, Associate Professor, Principal Investigator — Kahramanmaras Sutcu Imam University; Abdülkadir Ertürk, Msc, Principal Investigator — Kahramanmaras Sutcu Imam University; Yusuf Şinasi Kırmacı, Asisstant Prof, Study Chair — Kahramanmaras Sutcu Imam University; mehmet göğremiş, Asisstant Prof, Study Chair — Kahramanmaras Sutcu Imam University; Mehtap Sönmez, Professor, Study Chair — Kahramanmaras Sutcu Imam University; Suat Erel, Professor, Study Director — Pamukkale University; Emel Taşvuran Horata, Study Chair — Sakarya University of Applied Sciences
Locations (1):
- Kahramanmaraş Sütçü imam University, Faculty of Health Science, Department of Physiotherapy and Rehabilitation, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No